CLINICAL TRIAL: NCT04624854
Title: Dual Anti-Platelet Therapy in Patients With Coronary Multi-Vessel Disease (DAPT-MVD): A Prospective, Multicenter, Randomized, Controlled Trial
Brief Title: Dual Anti-Platelet Therapy in Patients With Coronary Multi-Vessel Disease (DAPT-MVD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Collaborators: Chinese Society of Cardiology (Other); Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yu Bo, Director, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAPT-MVD-201912
Record Dates: First submitted 2020-10-27; First posted 2020-11-12 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome; Heart Diseases; Syndrome Heart Disease; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Coronary Disease; Vascular Diseases
Keywords: Coronary multivessel disease; Dual antiplatelet therapy; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Coronary Disease; Vascular Diseases | interventions — Clopidogrel

STUDY DESIGN:
Intervention Model Description: All patients will be randomly divided into the treatment group and control group on a 1:1 basis, based on a permuted completely randomization. The treatment group will use aspirin + clopidogrel dual anti-platelet therapy for 12 months, and the control group will use aspirin monotherapy for 12 months.
Masking Description: This is an open-label trial, and the investigators and subjects will not be blinded. Under these conditions, the following methods will be employed to minimize bias:
  1. Clinical Endpoint Committee (CEC) is an independent group of experts that reviews clinical trial data in order to give expert opinions about clinical safety or efficacy events of interest;
  2. The statisticians are independent and blind to the grouping information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin monotherapy (Placebo Comparator): Patients will receive aspirin monotherapy without co-administration of clopidogrel for 12 months after randomization.
  Interventions: Drug: Aspirin monotherapy
- Clopidogrel and aspirin dual-antiplatelet therapy (Experimental): Patients will receive co-administration of clopidogrel and aspirin for 12 months after randomization.
  Interventions: Drug: Clopidogrel and aspirin dual-antiplatelet therapy

INTERVENTIONS:
Drug: Clopidogrel and aspirin dual-antiplatelet therapy — Patients will receive co-administration of clopidogrel and aspirin for 12 months after randomization.
  Arms: Clopidogrel and aspirin dual-antiplatelet therapy
Drug: Aspirin monotherapy — Patients will receive aspirin monotherapy without co-administration of clopidogrel for 12 months after randomization.
  Arms: Aspirin monotherapy

SUMMARY:
This study is a prospective, multicenter, parallel, open-label, randomized, controlled, superiority trial. It is planned to recruit 8,250 patients with multi-vessel disease(MVD), and the patients will be followed-up for at least 12 months after being implanted with a drug-eluting stent (DES) at one of 100 different centers. All patients will be randomly divided into the treatment group and control group on a 1:1 basis, based on a permuted completely randomization.

ELIGIBILITY:
Inclusion Criteria:

* The enrolled subjects must meet all of the following criteria:

  1. Aged 18-75 years old (inclusive).
  2. Patients with MVD who underwent DES implantation for 12 months.
  3. Patients have been treated with aspirin and can tolerant of aspirin at doses of 75-150 mg/day as maintenance therapy during the study period.
  4. Patients have signed informed consent.

Exclusion Criteria:

- Subjects who meet any one of the following criteria are excluded from the study:

1. Planned to use of ADP receptor blockers (eg, clopidogrel, ticagrelor, and ticlopidine), dipyridamole, or cilostazol.
2. Contraindication to ADP receptor blockers or aspirin.
3. Planned to use anticoagulants during the study period.
4. Planned coronary, cerebrovascular, or peripheral arterial revascularization during the study period.
5. Planned major cardiac or non-cardiac surgery during the study period.
6. Concomitant oral or intravenous therapy with CYP2C19 medium or strong inhibitors.
7. Known severe liver disease(ALT/AST is 3 times above normal).
8. Subjects with renal failure who required or anticipated dialysis during the study period.
9. Platelet count <50×10^9/L.
10. Patients with:

    * A history of intracranial bleed or ischemic stroke at any time.
    * A central nervous system tumor or intracranial vascular abnormality (eg, aneurysm, arteriovenous malformation) at any time.
    * Intracranial or spinal cord surgery within 5 years.
11. Pregnancy or lactation or planned to pregnant during the study period.
12. Life expectancy < 1 year.
13. Any condition which in the opinion of the investigator would make it unsafe or unsuitable for the patient to participate in this study (eg, active malignancy other than squamous cell or basal cell skin cancer).
14. Concern for inability of the patient to comply with study procedures and/or followup (eg, alcohol or drug abuse).
15. Participation in another clinical study and did not reach the major endpoint.
16. Involvement in the planning and/or conduct of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8250 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Incidence of MACCE(cardiovascular death, nonfatal myocardial infarction or nonfatal stroke). | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of MACCE in patients with MVD.

SECONDARY OUTCOMES:
Incidence of all-cause mortality. | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of all-cause mortality in patients with MVD.
Incidence of cardiovascular death. | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of cardiovascular death in patients with MVD.
Incidence of nonfatal myocardial infarction. | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of nonfatal myocardial infarction in patients with MVD.
Incidence of nonfatal stroke. | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of nonfatal stroke in patients with MVD.
Incidence of NACE (net adverse clinical events). | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of net adverse clinical events (MACCE and BARC type 2-5 bleeding) in patients with MVD.
Incidence of cardiovascular death or hospitalization. | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of cardiovascular death or hospitalization (myocardial infarction, stroke, emergency revascularization, unstable angina or TIA) caused by thrombotic events in patients with MVD.
Incidence of emergency revascularization. | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of emergency revascularization in patients with MVD.
Incidence of repeat revascularization. | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of any repeat revascularization in patients with MVD.
Incidence of definite/possible stent thrombosis. | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of definite/possible stent thrombosis in patients with MVD.

OTHER OUTCOMES:
Incidence of clinically relevant bleeding events. | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of clinically relevant bleeding events (BARC type 2-5 bleeding) in patients with MVD.
Incidence of major bleeding events. | Through study completion, median follow-up duration is 34.3 months.
  To evaluate the effect of clopidogrel and aspirin dual-antiplatelet therapy on the incidence of major bleeding events (BARC type 3-5 bleeding) in patients with MVD.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, M.D.,FACC, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (97):
- China (97):
  - Xinqiao Hospital, Army Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fuzhou University Affiliated Provincial Hospital, Fuzhou, Fujian
  - The Fifth Hospital of Xiamen, Xiamen, Fujian
  - Guangdong Provincial People's Hospital, Zhongshan, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Central South University Xiangya School of Medicine Affiliated Haikou Hospital, Haikou, Hainan
  - Hainan General Hospital (Hainan Affiliated Hospital of Hainan Medical University), Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Pingquan County Hospital, Chengde, Hebei
  - Harrison International Peace Hospital, Hengshui, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Shijiazhuang, Shijiazhuang, Hebei
  - Tangshan Central Hospital, Tangshan, Hebei
  - The Second Affiliated Hospital of Xingtai Medical College, Xingtai, Hebei
  - The Fifth Affiliated Hospital of Qiqihar Medical College, Daqing Longnan Hospital., Daqing, Heilongjiang
  - Daqing People's Hosipital, Daqing, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Hospital of Harbin, Harbin, Heilongjiang
  - Heilongjiang Provincial Hospital, Harbin, Heilongjiang
  - The Second Hospital of Harbin, Harbin, Heilongjiang
  - Harbin 242 Hospital, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Beidahuang Industry Group General Hospital, Harbin, Heilongjiang
  - Shuangcheng People's Hospital, Harbin, Heilongjiang
  - Hegang Hekuang Hospital, Hegang, Heilongjiang
  - People's Hospital of Hegang City, Hegang, Heilongjiang
  - The Baoquanling Hospital of Beidahuang Group, Hegang, Heilongjiang
  - Nenjiang People's Hospital, Heihe, Heilongjiang
  - Jiamusi Central Hospital, Jiamusi, Heilongjiang
  - The First Affiliated Hospital of Jiamusi University, Jiamusi, Heilongjiang
  - Jiansanjiang Hospital of Beidahuang Group, Jiamusi, Heilongjiang
  - Jixi Jikuang Hospital, Jixi, Heilongjiang
  - Jixi People's Hospital, Jixi, Heilongjiang
  - Mishan People's Hospital, Mishan, Heilongjiang
  - Mudanjiang City Second People's Hospital, Mudanjiang, Heilongjiang
  - Hongqi Hospital Affiliated to Mudanjiang Medical University, Mudanjiang, Heilongjiang
  - Mudanjiang Cardiovascular Hospital, Mudanjiang, Heilongjiang
  - Mudanjiang First People's Hospital, Mudanjiang, Heilongjiang
  - Mudanjiang Hospital of Beidahuang Group, Mudanjiang, Heilongjiang
  - Qiqihar Jianhua Hospital, Qiqihar, Heilongjiang
  - The Third Affiliated Hospital of Qiqihar Medical University, Qiqihar, Heilongjiang
  - The First Affiliated Hospital of Qiqihar Medical University, Qiqihar, Heilongjiang
  - Shuangyashan Mining Group Hospital, Shuangyashan, Heilongjiang
  - Shuangyashan People's Hospital, Shuangyashan, Heilongjiang
  - Baoqing County People's Hospital, Shuangyashan, Heilongjiang
  - The Hongxinglong Hospital of Beidahuang Group, Shuangyashan, Heilongjiang
  - The First Hospital of Suihua City, Suihua, Heilongjiang
  - People's Hospital of Daxing'anling Region, Xing'anling, Heilongjiang
  - Tieli Medical Service Community Central Hospital, Yichun, Heilongjiang
  - The First Hospital of Yichun City, Yichun, Heilongjiang
  - Yichun Forestry Central Hospital, Yichun, Heilongjiang
  - Kaifeng Central Hospital, Kaifeng, Henan
  - Nanyang First People's Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - Puyang People's Hospital, Puyang, Henan
  - First People's Hospital of Shangqiu, Shangqiu, Henan
  - Central Hospital of Yongcheng, Shangqiu, Henan
  - Xinxiang Second People's Hospital, Xinxiang, Henan
  - The People's Hospital of Yongcheng, Yongcheng, Henan
  - The 7th People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Dancheng County People's Hospital, Zhoukou, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - Hulunbuir People's Hospital, Hulunbuir, Inner Mongolia
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - Affiliated Pizhou Hospital of Xuzhou Medical University, Pizhou, Jiangsu
  - First People's Hospital of Fuzhou, Fuzhou, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Third Betune Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Jilin Central General Hospital, Jilin, Jilin
  - Jilin Hospital of Chinese and Western Medicine, Jilin, Jilin
  - Songyuan Central Hospital, Songyuan, Jilin
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Central Hospital of Dalian University of Technology (Dalian municipal central hospital ), Dalian, Liaoning
  - General Hospital of Ningxia Medical University - Cardiovascular and Cerebrovascular Hospital, Yinchuan, Ningxia
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Shandong Healthcare Group Feicheng Hospital, Feicheng, Shandong
  - The Fifth People's Hospital of Jinan, Jinan, Shandong
  - Shandong Second Provincial General Hospital, Jinan, Shandong
  - The Fourth People's Hospital of Jinan, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Second People's Hospital of Liaocheng, Liaocheng, Shandong
  - The Affiliated Taian City Centeral Hospital of Qingdao University, Tai’an, Shandong
  - Zhongshan Hospital Wusong Branch, Fudan University, Shanghai, Shanghai Municipality
  - Dazhou Central Hospital, Dazhou, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tian J, Wang Z, Wang Y, Wang F, Wang Y, Zhao P, Hou X, Peng X, Tian M, Wang D, Yu B. Rationale and Design of Dual Antiplatelet Therapy in Patients with Coronary Multi-Vessel Disease (DAPT-MVD): A Multicenter, Randomized, Controlled Trial. Clin Cardiol. 2024 Dec;47(12):e70049. doi: 10.1002/clc.70049. PMID 39587825